CLINICAL TRIAL: NCT04353180
Title: Isotretinoin in Treatment of COVID-19 (Randomized)
Brief Title: Assessment the Activity Value of Isotretinoin (13- Cis-Retinoic Acid ) in the Treatment of COVID-19 ( Isotretinoin in Treatment of COVID-19) (Randomized)
Acronym: Isotretinoin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Collaborators: The First Hospital of Jilin University (Other); 2-Montefiore Health System and Albert Einstein College of Medicine, Newyork, United States of America (U.S.A). (Unknown)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Sponser Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Proposed by Mahmoud Elkazzaz
Record Dates: First submitted 2020-04-10; First posted 2020-04-20 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: COVID19
Keywords: COVID 2019, ,T Cells, IFN type1; Retinoic acid; Endosomal toll-like receptor 3; T Cells; IFN type1; AT1; ACE2
MeSH Terms: conditions — COVID-19 | interventions — Isotretinoin; Capsules

STUDY DESIGN:
Intervention Model Description: Patients and method :
  This study will performed on 10000 patients tested positive for the presence of COVID-19 RNA by RT-PCR kit for RNA detection will randomly divided into 5 equal groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- 13 cis retinoic acid doses orally plus the standard therapy (Active Comparator): Arm 1: infected patients will receive the standard therapy for COVID-19 (Paracetamol 500 mg /6h, Hydroxychloroquine 500 mg/ 12h, Oseltamivir 150 mg /12 h for 5 days, Azithromycin 1 gm first day then 500 mg/day for 1st line or Clarithromycin 500 mg/12 h for 7-14 days, Ascorbic acid 500 mg/12 h and Cyanocobalamin IV once daily plus Lopinavir 400mg/Ritonavir 100 mg caps 2 capsules twice daily in severe cases) and after three days of the standard therapy the infected patients will receive 13 cis retinoic acid (0.5 mg/kg/day in 2 divided doses orally for 14 days combined with the standard therapy . All subjects were encouraged to complete the full course of treatment and common side effects were explained. Side effects and compliance will be documented.
  Interventions: Drug: Drug Isotretinoin (13 cis retinoic acid ) capsules+standard treatment
- Aerosolized 13 cis retinoic acid plus the standard therapy (Active Comparator): Arm 2: infected patients will receive the standard therapy for COVID-19 (Paracetamol 500 mg /6h, Hydroxychloroquine 500 mg/ 12h, Oseltamivir 150 mg /12 h for 5 days, Azithromycin 1 gm first day then 500 mg/day for 1st line or Clarithromycin 500 mg/12 h for 7-14 days, Ascorbic acid 500 mg/12 h and Cyanocobalamin IV once daily plus Lopinavir 400mg/Ritonavir 100 mg caps 2 capsules twice daily in severe cases) and after three days of the standard therapy the infected patients will receive Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days
  Interventions: Drug: Isotretinoin(Aerosolized 13 cis retinoic acid) +standard treatment
- 13 cis retinoic acid doses orally (Active Comparator): Infected patients will receive 13 cis retinoic acid (0.5 mg/kg/day in 2 divided doses orally for 14 days
  Interventions: Drug: Isotretinoin (13 cis retinoic acid ) capsules
- Aerosolized 13 cis retinoic acid (Active Comparator): The infected patients will receive Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days
  Interventions: Drug: Aerosolized 13 cis retinoic acid
- The standard therapy (Sham Comparator): Arm 3:infected patients will receive the standard therapy for COVID-19 for 14 days
  Interventions: Drug: Standard treatment

INTERVENTIONS:
Drug: Drug Isotretinoin (13 cis retinoic acid ) capsules+standard treatment — After three days of randomization and standard treatment , 13 cis retinoic acid (0.5 mg/kg/day in 2 divided doses orally for 14 days.+standard treatment
  Standard treatment is according to the protocol of treatment of 2019-nCoV infection
  Other Names: 13 cis retinoic acid
  Arms: 13 cis retinoic acid doses orally plus the standard therapy
Drug: Isotretinoin(Aerosolized 13 cis retinoic acid) +standard treatment — Drug: After three days of randomization and standard treatment , Aerosolized 13 cis retinoic acid in gradual two doses increase froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days +standard treatment
  Standard treatment is according to the protocol of treatment of 2019-nCoV infection
  Other Names: Aerosolized 13 cis retinoic acid
  Arms: Aerosolized 13 cis retinoic acid plus the standard therapy
Drug: Isotretinoin (13 cis retinoic acid ) capsules — 13 cis retinoic acid (0.5 mg/kg/day in 2 divided doses orally for 14 days
  Arms: 13 cis retinoic acid doses orally
Drug: Aerosolized 13 cis retinoic acid — Aerosolized 13 cis retinoic acid in gradual two doses increase froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days
  Arms: Aerosolized 13 cis retinoic acid
Drug: Standard treatment — Standard treatment is according to the protocol of treatment of 2019-nCoV infection
  Arms: The standard therapy

SUMMARY:
Assessment the Activity Value of Isotretinoin (13- Cis-Retinoic Acid ) in the Treatment of COVID-19

Mahmoud ELkazzaz(1),Tamer Haydara(2), Mohamed Abdelaal(3), Abedelaziz Elsayed(4) ,Yousry Abo-amer(5), Hesham Attia(6), Quan Liu(7)' Tim Duong(8) and Heba Sahyon(9)

1. Department of chemistry and biochemistry, Faculty of Science, Damietta University, Egypt.
2. Department of Internal Medicine, Faculty of Medicine, Kafrelsheikh University, Egypt
3. Department of Cardiothoracic Surgery, Faculty of Medicine, Kafrelsheikh University, Egypt
4. Department of Pharmaceutical Biotechnology, Faculty of Pharmacy, Tanta University, Egypt.
5. Hepatology,Gastroenterology and Infectious Diseases Department, Mahala Hepatology Teaching Hospital, Egypt
6. Department of Immunology and Parasitology, Faculty of Science, Cairo University, Egypt.
7. School of Life Sciences and Engineering, Foshan University, Laboratory of Emerging Infectious Disease, Institute of Translational Medicine, The First Hospital of Jilin University, Changchun, China.
8. Montefiore Health System and Albert Einstein College of Medicine, New York, United States of America.
9. Chemistry Department, Faculty of Science, Kafrelsheikh University, Egypt.

   * This clinical study is the first clinical study in literature (submitted on 20 April, 2020) which demonstrated that Isotretinoin will provide complete protection against COVID-19

Abstract

The COVID-19 pandemic caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has infected over 100 million people causing over 2.4 million deaths over the world, and it is still expanding. There is an urgent need for targeted and effective COVID-19 treatments which has put great pressure on researchers across the world for developing effective drugs. In this clinical study we attempt to demonstrate Isotretinoin could be an effective and promising treatment for SARS-CoV-2 based on the intracellular mechanism of SARS-CoV-2 transmission and consequences caused. Isotretinoin could strongly inhibit both inflammation and viral entry in severe acute respiratory syndrome coronavirus 2 infection via decreasing the overproduction of early response proinflammatory cytokines (interleukin-6 ) which are over expressed in COVID-19 and contributed to disease progression, poor outcomes, vascular hyper permeability and multiorgan failure in patients infected with COVID-19. It could also block the entry of COVID-19 by inhibiting androgenic factors that induce serine 2 transmembrane protease (TMPRSS2) expressions.. In addition to inhibiting of Angiotensin-converting enzyme-2 (ACE2), Angiotensin T1 protein and Angiotensin II-mediated intracellular calcium release pathway which is responsible for COVID-19 cell fusion and entry, ACE2-expressing cells are prone to SARS-CoV-2 infection as ACE2 receptor facilitates cellular viral entry and invasion. Moreover, isotretinoin is a potential repressor and inhibitor of papain-like protease (PLpro), which is a lethal protein expressed by COVID-19 genes and is an enzyme of dubiquitination which facilitates virus replication in patients with COVID-19.The genome of Middle East Respiratory Syndrome Coronavirus is recognized by melanoma differentiation-associated protein-5 (MDA5), retinoic acid inducible gene-1 (RIG-1) and endosomal toll-like receptor 3 (TLR3) as pathogen-associated molecular patterns. This recognition resulted in the formation of type-1 interferon (IFN1). As an evasion mechanism, virus synthesize proteins that hinder the production IFN1 in the pathway. 13-cis retinoic acid induced significant upregulation of toll-like receptor 3 (TLR3), mitochondrial antiviral-signaling protein (MAVS) and IFN regulatory factor 1 expression in a time-dependent. Furthermore, 13 cis Retinoic Acid (13 cis RA) could be an effective and promising treatment for SARS-CoV-2 owing to its ability to increase CD4 cells and induce mucosal IgA antibodies that are less prone to Antibody Dependent Enhancement process (ADE) and responsible for passive mucosal immunity in the respiratory tract. ADE is a phenomenon in which antiviral antibodies facilitate viral infection of target immune cells and, in some cases, make a second infection worse, such as dengue fever (dengue virus), By inducing IgA antibodies, 13 cis retinoic acid enhances mucosal immunity and is known to be a potent IgA isotype.13 Cis retinoic acid induced significant upregulation of toll-like receptor 3 an immune boosting action that may result in an immune response to dsRNA intermediate leading to the production of type I IFNs which is important to enhance the release of antiviral proteins for the protection of uninfected cells. Isotretinoin therapy has furthermore proven anti-platelet and fibrinolytic activities which may protect patients infected with covid-19 from widespread blood clots. From this point, we suggest that isotretinon will be the Immunity passport" in the context of COVID-19

DETAILED DESCRIPTION:
The study is a randomized interventional comparative Phase III trial. 10000 adult male and female patients with positive COVID-19 diagnosis and fulfilling the below outlined inclusion criteria will be enrolled into the study.

Isotretinoin(13cis RA) may be able to inhibit COVID 2019 entry via down regulation of ACE2 , AT1 protein and Ang II-mediated intracellular calcium release rather than inhibition of interleukin-6 (IL-6) and this is discussed as follow :

The COVID-19 pandemic caused by SARS-COV-2 has infected over 2,000,000 people causing over 150,000 deaths. A key host cellular protein required for the virus entry is angiotensin-converting enzyme 2 (ACE2) whose expression has been demonstrated in many tissues including alveolar epithelial type II cells in lungs, oral mucosa ,intestine, heart, kidney, endothelium and skin. ACE2-expressing cells can act as home cells and are prone to SARS-CoV-2 infection as ACE2 receptor facilitates cellular viral entry and replication. A study demonestrated that patients with hypertension and diabetes mellitus may be at higher risk of SARS-CoV-2 infection, as these patients are often treated with ACE inhibitors (ACEIs) or angiotensin II type-I receptor blockers (ARBs), which have been previously suggested to increase ACE2 expression. In another study by Sinha et al who analyzed a publicly available Connectivity Map (CMAP) dataset of pre/post transcriptomic profiles for drug treatment in cell lines for over 20,000 small molecules, isotretinoin was the strongest down-regulator of ACE 2 receptors. On the other hand, they found 6 drugs in CMAP that are currently being investigated in clinical trials for treating COVID-19 (chloroquine, thalidomide, methylprednisolone, losartan, lopinavir and ritonavir, from clinicaltrials.gov), none of which was found to significantly alter ACE2 expression (P>0.1) Moreover, another study demonstrated that isotretinoin is a potential papain like protease (PLpro) inhibitor which is a protein encoded by SARS-CoV-2 genes and considered one of the proteins that should be targeted in COVID-19 treatment by performing target-based virtual ligand screening.

Previous studies on the related severe acute respiratory syndrome coronavirus (SARS-CoV) and SARS-CoV FP FP have shown that calcium (Ca2+) plays an important role for fusogenic activity via a Ca2+ binding pocket with conserved glutamic acid (E) and aspartic acid (D) residuesdemonstrated that intracellular Ca2+ enhances MERS-CoV WT PPs infection by approximately two-fold and that E891 is a crucial residue for Ca2+interaction. Electron spin resonance revealed that this enhancement could be attributed to Ca2+ increasing MERS-CoV FP fusion-relevant membrane ordering. Intriguingly, isothermal calorimetry titration showed that MERS-CoV FP binds one Ca2+, as opposed to SARS-CoV FP which binds to two Ca2+ ion.

Angiotensin II increases the intracellular calcium activity in podocytes of the intact glomerulus. The L-type Ca2+ channel blocker nicardipine did not influence the Ang II-mediated [Ca2+] increase and it has been postulated that SARS-CoV-2 binding to ACE2 may attenuate residual ACE2 activity, skewing the ACE/ACE2 balance to a state of heightened angiotensin II activity leading to pulmonary vasoconstriction and inflammatory and oxidative organ damage, which increases the risk for acute lung injury (ALI). AngII via AT1 receptors upregulates many proinflammatory genes, such as vascular cell adhesion molecule-1 (VCAM-1), intercellular adhesion molecule-1 (ICAM-1), interleukin-6 (IL-6).30 but 13cis RA specifically down-regulated the AT1 protein in a dose- and time-dependent manner. Down-regulation of the AT1 expression leads to reduced AngII-mediated intracellular calcium release Similarly with receptor down-regulation, Treatment with 13cRA resulted in a significant reduction in AT1 mRNA .13cRA has a glucose- and RAR/RXR independent mechanism for transcriptional inhibition of AT1,

Isotretinoin(13cis RA) and ATRA may be able to inhibit COVID 2019 infection via inducing the antiviral immunity and this is discussed as follow :

Since effective immune response against viral infections depends on the activation of cytotoxic T cells that can clear infection by killing virus-infected cells , boosting the numbers and function of T cells in COVID-19 patients is critical for successful recovery. A recent study reported that the 82.1% of COVID-19 cases displayed low circulating lymphocyte counts. A CoV infects macrophages, and then macrophages present CoV antigens to T cells. This process leads to T cell activation and differentiation, including the production of cytokines associated with the different T cell subsets (Th17), followed by a massive release of cytokines for immune response amplification. The continued production of these mediators due to viral persistence has a negative effect on NK, and CD8 T cell activation. However, CD8 T cells produce very effective mediators to clear CoV However, the factors which might cause the reduction in count, and the activation status of T cells in COVID-19 patients, remain uninvestigated.

Recent study of 522 COVID patients and 40 healthy controls from two hospitals in Wuhan, China demonstrated that T cell numbers are negatively correlated to serum IL-6, IL-10 and TNF-α concentration, with patients in decline period showing reduced IL-6, IL-10 and TNF-α concentrations and restored T cell counts. T cells from COVID-19 patients have significantly higher levels of the exhausted marker programmed cell death protein(PD-1) as compared to health controls. Moreover, increasing PD-1 and Tim-3 expression on T cells could be seen as patients progressed from prodromal to overtly symptomatic stages, further indicative of T cell exhaustion. T cell exhaustion is a progressive loss of effector function due to prolonged antigen stimulation, characteristic of chronic infections. Dendritic cell inhibition is connected to exhaustion of CD8+ T cell polyfunctionality during chronic hepatitis C virus infection. CD8 T cells produce very effective mediators to clear nCoV2019.

Dendritic cells (DCs) play a key role in innate immune and adaptive immune responses. As the strongest antigen presenting cells in the organism, they effectively stimulate the activation of T lymphocytes and B lymphocytes, thus combining innate and adaptive immunity. Immature DCs have strong migration ability, and mature DCs can effectively activate T cells in the central link of startup, regulation, and maintenance of immune responses. Thus, once the maturation process of DCs is blocked, it directly affects the initiation of subsequent adaptive immune response. MERS-CoV-2 is able to affect human dendritic cells and macrophages in-vitro .Productive replication of Middle East respiratory syndrome coronavirus in monocyte-derived dendritic cells modulates innate immune response.

Another study proposed that C -C chemokine receptor type 4 (CCR4) contributes to T cell lung homing imprinting. It was found that lung DCs induce the expression of CCR4 on T cells. Lung DCs-activated T cells traffic more efficiently into the lung and protect against influenza more effectively compared with T cells activated by DCs from other tissues. Lim and colleagues suggested that CXCR4 plays a role in CD8+ T cell migration to airway tissues

Dendritic cell inhibition is connected to exhaustion of CD8+ T cell polyfunctionality during chronic hepatitis C virus infection. CD8 T cells produce very effective mediators to clear nCoV2019

Presence of RA in different tissues is very imprtant for immune induction and fighting viral infection, for example, RA is present at high concentrations in the small intestine due to metabolizing dietary vitamin A by gut epithelial cells. In this local environment, RA activates and primes dendritic cells (DCs) to become CD103+ DCs that produce RA.3, 4CD103+ DCs are migratory cells that activate naive T cells in mesenteric lymph nodes to become effector T cells that contribute to both intestinal homeostasis and immunity.and also RA is an important signal that induces IgA-producing B cells. The gut homing T cells and B cells play essential roles in protecting the digestive tract from pathogens.

Retinoic acid (atRA) can inhibit the spontaneous apoptosis of activated human T lymphocytes in vitro. 13-cis RA activates Th2 cytokine production Enhanced circulating dendritic cell numbers.

So, according to this previous studies the principal investigator suggests that T cells lymphopenia and exhaustion may be resulted by Dendritic cells (DCs) infection and inhibition by MERS-CoV-2.

Retinoic acid has profound effects on cellular proliferation and differentiation. Moreover, it has been reported that ATRA exhibits both anti-inflammatory and immunoregulatory effects. Recent studies have shown that FOXP3 expression and the immune function of Regulatory T cells (Tregs ) can be enhanced by ATRA in in both patients and mouse models. .13Retinoic acid (RA) is produced by a number of cell types, including macrophages and dendritic cells, which express retinal dehydrogenases that convert vitamin A to its main biologically active metabolite, all-trans RA. All-trans RA binds to its nuclear retinoic acid receptors that are expressed in lymphoid cells and act as transcription factors to regulate cell homing and differentiation. RA production by CD103+ dendritic cells and alveolar macrophages functions with TGF-b to promote conversion of naive T cells into Foxp3+ regulatory T cells and, Thereby, maintain mucosal tolerance

So, principal investigator expects high inducing of Dendritic cells (DCs) by retinoic acid treatment which will lead to T cells activation and migration with less exhaustion phenomenon.

According to this protocol treatment with retinoic acid will induce FOXP3 and CD8+,CD4+,CD25+,FOXP3+ Tregs which their absence during acute infection alters the ability of the host to limit tissue damage and inducesT cells which were dramatically reduced in COVID-19 patients to exert its antiviral and anti-inflammatory effect protecting lung cells and neural cells from the inflammatory and the destructive effect of IL-6, IL-1, and TNF-α which are induced and highly expressed in COVID 2019 patients.

Researchers from Wenzhou, China looked at clinical laboratory features including lipid levels of patients with COVID 19. They found dramatic reductions in the cholesterol levels of patients infected with COVID 19, compared with healthy controls .The study provides data to suggest that cholesterol levels decline quite rapidly during the early stages of infection and increase as the patient starts to recover. Therefore, indicating that cholesterol may have an important role to play in defending the body against such infections According to our protocol depending on previous studies the principal investigator demonstrated that there is a strong relation between immune system and cholesterol levels .When the cholesterol level is low specifically in the case of viral infection like COVID 2019 infection the immune system is impaired and the antiviral immune cells will be declined and inhibited :-

Cellular cholesterol is a component of the plasma membrane and is also essential in cell proliferation. Regulation of intracellular cholesterol levels has been proposed as a mechanism to regulate T cell and macrophages proliferation. Intracellular cholesterol level is regulated by two competing pathways, cholesterol uptake and efflux, and ABCA1 plays a major role in the cholesterol efflux pathway. The ATRA induces ABCA1 expression and ABCA1-dependent cholesterol efflux in activated primary human CD4+ T cells implying that RA could affect T cell functions by regulating the cellular cholesterol levels.

ATRA upregulates ABCA1 expression only in activated CD4+ T cells, indicating that induction of ABCA1 by ATRA and 13 cis Retinoic Acid may play an important role in immune response.

Retinoic acid and liver X receptor agonist synergistically inhibit HIV infection in CD4+ T cells by up-regulating ABCA1-mediated cholesterol efflux.

So, the principal investigator expects that retinoic acid treatment will highly induce T cells and anti-inflammatory regulatory T cells, T helper via cholesterol efflux and inducing ATP-binding cassette transporter (ABCA1) and protect lung and neural cells and inhibit COVID 2019 infection.

The genome of Middle East Respiratory Syndrome Coronavirus is recognized by melanoma differentiation-associated protein-5 (MDA5), retinoic acid inducible gene-1 (RIG-1) and endosomal toll-like receptor 3 (TLR3) as pathogen-associated molecular patterns. This recognition resulted in the formation of type-1 interferon (IFN1). As an evasion mechanism, virus synthesize proteins that hinder the production IFN1 in the pathway.

RA also acts directly on macrophages at both mucosal sites and other immunological sites. AtRA modulates peritoneal macrophage activation by endotoxin and IFN-γ by suppressing TNF production and nitric oxide (NO) synthesis .In addition, at RA inhibits the expression of PGE2 and COX-2 and the release of TNF, which are induced by bacterial lipopolysaccharide (LPS) in murine peritoneal macrophages .

A study reported recently that substance (ATRA) have preventive effects on pulmonary fibrosis by inhibiting IL-6-dependent proliferation and TGF-β1-dependent trans differentiation of lung fibroblasts. Also, another studies demonstrated that 13-cis-retinoic acid and other retinoid analogs inhibit IL-1-induced IL-6 production and that this effect is analog-specific and, at least partially, transcriptionally mediated. This effect was dose-dependent with an IC50 of 10(-7) M RA and significant inhibition being noted with doses of RA as low as 10(-8) M. IL-10 production was inhibited by ATRA administration.

A study demonstrated that TLR3(-/-), TLR4(-/-), and TRAM(-/-) mice are more susceptible to SARS-CoV than wild-type mice but experience only transient weight loss with no mortality in response to infection. In contrast, mice deficient in the TLR3/TLR4 adaptor TRIF are highly susceptible to SARS-CoV infection, showing increased weight loss, mortality, reduced lung function, increased lung pathology, and higher viral titers . New studies showed that the high level of IFN-α/β produced from the TLR3-IRF3/IRF7 pathway and IFN-β is the reason for inhibiting DENV replication. 13Cis retinoic Acid induced significant upregulation of toll-like receptor 3 (TLR3) resulting in an immune response to dsRNA intermediate which can be partially generated during CoV-2 replicationTLR3 sensitized by dsRNA and cascades of signaling pathways (IRFs and NFκB activation, respectively) are activated to produce type I IFNs. The production of type I IFNs is important to enhance the release of antiviral proteins for the protection of uninfected cells. Sometimes, accessory proteins of CoV can interfere with TLR3 signaling and bind the dsRNA of CoV during replication to prevent TLR3 activation and evade the immune response. 13Cis retinoic Acid induced significant upregulation of toll-like receptor 3 (TLR3) , mitochondrial antiviral-signaling protein (MAVS) and retinoid-induced gene I (RIG-I) and IFN regulatory factor 1 expression in a time-dependent.

In further research, Tsai .and Chen showed the high level of IFN-α/β produced from the TLR3-IRF3/IRF7 pathway and IFN-β is the reason for inhibiting DENV replication. In HUH-7 cells, huTLR3 can recognize DENV-1 and induce the expression of IFN-β, which can enhance the expression of huTLR3 on the contrary . TLR3 also induces type I IFN during WNV.

Doctors treating the sickest Covid-19 patients have zeroed in on a new phenomenon: Some people have developed widespread blood clots, their lungs peppered with tiny blockages that prevent oxygen from pumping into the bloodstream and body.As with so much else about the Covid-19 response, health experts are learning about the symptom on the fly. Blood clots are common in patients who are immobilized, but they seem to be smaller and cause far more severe damage in some Covid-19 patients. Doctors have said they see patients with blood clots forming not only in their lungs, but also in blood vessels. Autopsies have also revealed blood clots in kidneys and other organs, which some experts say suggests an overwhelming immune system response to the virus that inflicts harm on the body

Retinoic acid, is known to possess in vivo anti-inflammatory, anti-platelet and fibrinolytic activities. A study investigated the in vitro thrombin and platelet aggregation inhibitory activities of retinoic acid and retinaldehyde.Retinoic acid, retinaldehyde and retinol exhibited potent inhibition of thrombin, with IC50 values of 67μg/ml, 74μg/ml and 152μg/ml, respectively for the inhibition of thrombin (Sigma); and 49μg/ml, 74μg/ml and 178μg/ml, respectively for the inhibition of thrombin (plasma). Amongst vitamin A and its derivatives, retinoic acid showed the highest inhibition of both the forms of thrombin.

Isotretinoin(13cis RA) may be able to inhibit COVID 2019 infection via reversIing the androgenic induction and activation effect of (DHT) on TMPRSS2 expression and helps to prevent cleaving and activating both the spike protein (S) of COVID 2019 and the viral receptor, and this is discussed as follow :

TMPRSS2 is both the most frequently altered gene in primary prostate cancer and a critical factor enabling cellular infection by coronaviruses, including SARS-CoV-2. The modulation of its expression by steroids could contribute to the male predominance of severe infections and given that TMPRSS2 has no known indispensable functions, and inhibitors are available, it is an appealing target for prevention or treatment of respiratory viral infections

TMPRSS2, a key regulator in prostate cancerTMPRSS2 was first identified in prostate cancer shortly after the gene had been originally cloned. Prostate cancer cell lines strongly upregulated TMPRSS2 expression in response to androgens . TMPRSS2 is expressed on the luminal side of the prostate epithelium, and its expression is increased in prostate cancer tissue compared to non-cancerous prostate tissue. Notably, the TMPRSS2 gene is a partner in one of the most common gene fusion eventsin solid tumors: somatic gene rearrangements involving TMPRSS2 witha member of the ETS family of oncogenic transcription factors, most commonly ERG. This fusion occurs in approximately 50% of primary prostate cancers among men of European ancestry.While ERG is not normally regulated by androgen, the gene fusion juxtaposes the androgen receptor regulatory elements of TMPRSS2 with the ERG gene. The ERG gene is consequently controlled by androgen receptor signaling and expressed highly in prostate cancers harboring the TMPRSS2: ERG fusion. Intriguingly, the prevalence of the TMPRSS2: ERG fusion is lower in prostate tumors of both black and Asian men. The relevance of this to the current COVID-19 pandemic is unclear.TMPRSS2: ERG fusion- cancers also have a distinct set of risk factors related to hormonal signaling. For example, men with higher genetically determined transcriptional activity of the androgen receptor have a higher risk of TMPRSS2: ERG fusion-positive prostate cancer but not of fusion-negative prostate cancer

TMPRSS2 is an androgen receptor signaling target gene and an androgen-regulated cell-surface serine protease expressed predominantly in prostate and lung epithelial cell TMPRSS2 is normally expressed several fold higher in the prostate relative to any other human tissue, though the normal physiological function(s) remains unknown. Importantly, unlike other TTSPs, TMPRSS2 transcription is regulated by androgenic ligands and the androgen receptor (AR). There is a positive correlation between AR and TMPRSS2 in microdissected primary tumor epithelium (r2 = 0.39 ; p <0.001).

Dihydrotestosterone (DHT) significantly and dramatically induced the expression of TMPRSS2 protein with two molecular masses of 60 (full-length) and 38 kDa (N-terminus) in a dose responsive manner

Data from Chinese outbreak show death rates for men almost 50 per cent higher than for women show that Early research from China suggests women and children are less likely to die than men if they catch the coronavirus. Death rates for Covid-19, the disease those infected with the coronavirus develop, are low for everyone: only 2.4 per cent of the 44,672 people in the Chinese study died. But although roughly even numbers of men and women catch the disease, men are more likely to develop such a serious case of Covid-19 they die.

More than 70 percent of Italy's coronavirus deaths have been among men but scientists there admit they are mystified by the gender gap. At least 3,400 people in Italy have died of the devastating disease - it yesterday announced it had a higher death Toll than China - but less than 1,000 of them have been women. Men are also more likely to pick up the infection in the first place and account for 60 percent of confirmed cases, according to Italy's public health research agency. An earlier analysis found that 80 per cent of the deaths were in men and just 20 per cent were in women - but the gap has narrowed over time

According to this data the principal investigator thinks that there is a strong relation between high mortality in males and androgenic effect specifically the effect of DHT on TMPRSS2 protein which is used by covid 2019 in cell invasion and entry and depending on this data related to six hormones specifically (DHT) , The investigator was able to discover whey women and children less likely to die from illness than men. So, the investigator divided infected patients according to their six hormone because TMPRSS2 is an androgen-regulated cell-surface serine protease expressed predominantly in prostate and lung epithelial cell TMPRSS2.

Androgen(DHT) potential effect on TMPRSS2 expression in children is less than its effect in females and males followed by viral severity and vigrousity in men compared with children and women. .

Androgen (DHT) potential effect on TMPRSS2 expression in females is less than in males followed by viral severity and vigrousity in men compared with females .

So, the principal investigator thinks that when some researchers investigated the role of sex steroids in SARS-CoV pathogenesis by comparing gonadectomized and control counterparts after infection. Gonadectomy or treatment with flutamide, a non-steroidal anti-androgen did not affect morbidity and mortality in male mice following lethal MA15 infection, They may be were wrong in their conclusions in suggesting that androgens do not play a role in SARS-CoV pathogenesis because Gonadectomy or treatment with flutamide will not completely affect or inhibit DHT and its derivatives(5α-Androstan-3α,17β-Diol) concentration in tissues and blood because after inhibiting testosterone with flutamide . the pathway of DHT formation will be activated to compensate the inhibited testosterone levels so the TMPRSS2 expression will be significantly induced by DHT and the treated animals will not be affected in case of flutamide treatment but in case of Gonadectomy the expression of TMPRSS2 will be decreased by DHT inhibition only if along time has passed on Gonadectomy in order to make sure that DHT and its derivatives completely declined in levels that will not allow it to affect on expression of TMPRSS2 and in female mice after blocking estrogen receptors it died because increasing formation of androgenic hormones.

A study demonstrated that 13- cis -Retinoic acid competitively and reversibly inhibits Dihydrotestosterone So, the principal investigator expects a significant modulation of TMPRSS2 expression after treating with 13- cis -Retinoic acid via temporary preventing the effect of dihydrotestosterone(DHT) on TMPRSS2 promoting and expression. And the type II transmembrane serine proteases TMPRSS2 which can cleave and activate the spike protein (S) of the severe acute respiratory syndrome coronavirus (SARS-CoV) for membrane fusion. In addition, these proteases cleave the viral receptor, the carboxypeptidase angiotensin-converting enzyme 2 (ACE2), and it was proposed that ACE2 cleavage augments viral infectivity.

A study demonstrated that COVID-19 reduces testosterone levels in men by altering the functioning of the gonads. So could the increased severity of the disease in men be due to lowered testosterone. But according to the principal investigator explanation COVID-19 reduces testosterone levels because there is a dramatic reductions in the cholesterol levels of patients infected with COVID 19, compared with healthy controls . Cholesterol levels decline quite rapidly during the early stages of infection and increase as the patient starts to recover.Therefore, indicating that cholesterol may have an important role to play in defending the body against such infections and depending on the principal investigator explanation, Testosterone is synthesized starting from cholesterol through a well-characterized steroid biosynthetic pathway involving the sequential action of multiple enzymes So, when cholesterol levels are decreased, this decrease will followed by decreasing in testosterone level and according to this explanation testosterone therapy in COVID 2019 is not recommended but temporary inhibitor of DHT is recommended such as Isotretinoin because this treatment by testosterone will inhibit cholesterol synthesis by feedback inhibition and decrease cholesterol uptake by Leydig cells in testis and this also will lead to over increase in DHT lvels and its derivatives in different tissues, which will induce TMPRSS2. because DHT is a potent activator of TMPRSS2 and this will be followed by processing and activation of COVID2019 spike protein to bined its ACE2 receptors in lung and kidney leading to their damage specifically in testis because it contains high levels of proteases and ACE2. Serine proteases are emerging as important contributors to the production, maturation, and functional competence of spermatozoa.

Depending on this data and according to this protocol, The principal investigator expects and suggests that retinoic acid is specific modulator of androgens specifically DHT not testosterone and could reverse the androgenic induction and activation effect of (DHT) on TMPRSS2 expression and prevent cleaving and activating both the spike protein (S) of COVID 2019 and the viral receptor, the carboxypeptidase angiotensin-converting enzyme 2 (ACE2). (All ideas and michanisms specifically role of Androgen in TMPRSS2 activation in COVID-19: Serendipity or opportunity for intervention and the inhibition of ACE2 ,AT1 protein and Ang II-mediated intracellular calcium release pathway which is responsible for SARS-CoV-2 cell fusion and entry included in the research protocol were submitted to Academy of scientific research and technology - Egypt- on 1 April , 2020. in Call no. 2/2019/ASRT- Ideation Fund)

________________________________________________________________________________________________________________________________________________________________________

Promising features of COVID 2019 treatment according Principal Investigator Protocol:

1. This medication have the feature of Aerosolized Drug Delivery to increase its efficacy beside Oral administration, Which makes it distinct from other medication in which should dose be only given orally. A study demonstrated that treating with 13 cis retinoic acid aerosolized via inhalation rout did not cause any damage in lung cells. Repeated high doses of 13 cis retinoic by inhalation resulted in moderate loss of body weight, but microscopic investigation of ten tissues including lung and oesophagus did not detect any significant aerosol-induced damage. The results suggest that administration of isotretinoin via powder aerosol inhalation is probably superior to its application via the oral route in terms of achieving efficacious drug concentrations in the lung.
2. Inhaled isotretinoin might provide sufficient drug to the target cells for efficacy while avoiding systemic toxicity.
3. A study demonstrated that 13 cis retinoic is used in treating Emphysema (emphysema is a lung condition that causes shortness of breath)
4. ATRA has been reported to induce formation of new alveoli and returns elastic recoil in the lung to approximately normal values in animal models of emphysema.
5. Strong expectation of complete COVID 2019 blockade from cell entry and infection depending on strong ethics, researches and references.
6. Availability of our compounds.
7. Ease of application.
8. Expectation of COVID 2019 treating of by more than one distinct mechanism.
9. Expectation of High induction of anti- inflammatory T cells and significant inhibition of IL-6 at low concentrations.
10. Controlling Accompanying cytokine storm.
11. No interactions with Egyptian protocol drugs were found.

ELIGIBILITY:
Inclusion Criteria:

Adult SARI patients with 2019-ncov infection confirmed by PCR; Absolute value of lymphocytes < 0. 6x 109/L; Severe respiratory failure within 48 hours and requires admission to ICU. (severe respiratory failure was defined as PaO2/FiO2 < 200 mmHg and was supported by positive pressure mechanical ventilation (including non-invasive and invasive mechanical ventilation, PEEP>=5cmH2O))

Exclusion Criteria:

Age < 18 Pregnant Allergic to experimental drugs and patients have the following conditions:

1. Hypercholesterolemia
2. Hypertriglyceridemia
3. Liver disease
4. Renal disease
5. Sjögren syndrome
6. Pregnancy
7. Lactation
8. Depressive disorder
9. Body mass index less than 18 points or higher than 25 points
10. Contraindications for hormonal contraception or intrauterine device.
11. Autoimmune diseases A history of organ, bone marrow or hematopoietic stem cell transplantation
12. Patients receiving anti-hcv treatment
13. Permanent blindness in one eye
14. History of iritis, endophthalmitis, scleral inflammation or retinitis 15-90 days of retinal detachment or eye surgery

16-The competent physician considered it inappropriate to participate in the study

------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------

Safety and promising features of isotretinoin in tne era of COVID 2019 according Principal Investigator Protocol:

1. This medication have the feature of Aerosolized Drug Delivery to increase its efficacy beside Oral administration, Which makes it distinct from other medication in which should dose be only given orally. A study demonstrated that treating with 13 cis retinoic acid aerosolized via inhalation rout did not cause any damage in lung cells.
2. Repeated high doses of 13 cis retinoic by inhalation resulted in moderate loss of body weight, but microscopic investigation of ten tissues including lung and oesophagus did not detect any significant aerosol-induced damage. The results suggest that administration of isotretinoin via powder aerosol inhalation is probably superior to its application via the oral route in terms of achieving efficacious drug concentrations in the lung.
3. Inhaled isotretinoin might provide sufficient drug to the target cells for efficacy while avoiding systemic toxicity.
4. A study demonstrated that 13 cis retinoic is used in treating Emphysema (emphysema is a lung condition that causes shortness of breath)
5. RA has been reported to induce formation of new alveoli and returns elastic recoil in the lung to approximately normal values in animal models of emphysema.
6. Strong expectation of complete COVID -19 blockade from cell entry and infection depending on strong ethics, researches and references.
7. Availability of our compounds.
8. Ease of application.
9. Expectation of COVID -19 treating by isotretinoin via more than one distinct mechanism.
10. Expectation of High induction of anti- inflammatory T cells and significant inhibition of IL-6 at low concentrations of isotretinoin.
11. Controlling Accompanying cytokine storm.
12. No interactions with Egyptian protocol drugs were found.
13. (13- cis -Retinoic acid ) can be given in the form of aerosol to avoid these systemic side effects. A clinical trial conducted on 148 subject from 5 university hospitals to evaluate the possibility of retinoids in the treatment of emphysema. The patients, were randomized to receive 13-cis retinoic acid (1 mg/kg/day, daily or ATRA at either low dose (1 mg/kg/day for 4 days/wk) or high dose (2 mg/kg/day for 4 days/wk), placebo for six months, followed by a three-month crossover phase. then, they were observed for an additional nine months before the final evaluation. In the trial, retinoids(13 cis retinoic acid ) were proven to be safe as the drug-related AEs were generally mild[188]. A study reported that the application of aerosolized RA system led to a rise of RA levels in lung, but not plasma. or liver. In lung concentration and levels of retinol, retinyl palmitate and retinyl stearate also showed to be unchanged [189] A study on rabbits demonstrated that 13 cis retinoic acid can be given in the form of aerosol without serious side effects In this study repeated elevated doses of 13 cis retinoic acid by inhalation caused moderate loss of body weight, but microscopic examination of ten tissues including oesophagus and lung did not found any significant inhalation-induced injury or damage therefore aerosolized 13 cis retinoic acid might provide sufficient therapy to the target cells in lung for efficacy while avoiding systemic toxicity © 2000 Cancer Research Campaign[190]

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
lung injury score | at 7and 14 days
  Proportion of lung injury score decreased or increased after treatment

SECONDARY OUTCOMES:
Absolute lymphocyte counts (CD4,CD8 and CD25+FOXP3+ Regulatory T) | at day 7 and 14 after randimization
Serum levels of IL-6,TNF,TLR3,CRP, ESR and Type I interferon | at day 7 and 14 after randimization
Serum level of COVID19 RNA | at day 7 and 14
  Serum level of COVID19 RNA
All cause mortality rate | at day 7 and 14
  died
Ventilation free days | at 14 days
  ventilation free days
ICU free days | at 14 days
  ICU free days
d-dimers | at 3-5days
  less than 250 ng/mL, or less than 0.4 mcg/mL of blood sample
Time to first negative SARS-CoV-2 PCR in NP swap | within 14 days
  (if pos. at baseline)
Angiotensin 1-7 (Ang 1-7) changes over time | at day 7 and 14
Angiotensin 1-5 (Ang 1-5) changes over time | at day 7 and 14
Renin changes over time | at day 7 and 14
Aldosterone changes over time | at day 7 and 14
Angiotensin-converting enzyme II (ACE2) changes over time | at day 7 and 14
Frequency of adverse events and severe adverse events | 14 days
Angiotensin II (Ang II) changes over time | at day 7 and 14
Sequential organ failure assessment score(SOFA score) over time | at day 7 and 14
Transe membrane protease ,serine II (TMPRSS2) changes over time | at day 7 and 14
Testosterone levels changes over time | at day 7 and 14
Dihydrotestosterone(DHT) levels changes over time | at day 7 and 14
Cholesterol levels changes over time | at day 7 and 14
Thrombin time (TT) | at day 7 and 14
IgA antibodies | at day 7 and 14
Melanoma differentiation-associated protein-5, retinoic acid inducible gene-1 (RIG-1) | at day 7 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Elkazzaz, B.Sc in Biochemistry, Principal Investigator — Faculty of Science, Damietta University; Dr.Tamer Hydara, Ass. Prof of Gastroenterology, Study Chair — Faculty of medicine kafr elshiekh university
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Kafr El-sheikh University, Cairo, Kafr el-Sheikh Governorate
  - Faculty of Medicine, Kafr El-sheikh University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided